CLINICAL TRIAL: NCT03825393
Title: Association of Ferritin Levels With Clinical Parameters in Patients With Fibromyalgia Syndrome
Status: Completed | Type: Observational
Sponsor: Tokat State Hospital (Other Government)
Responsible Party: Principal Investigator, Sevil Okan, principal investigator, Tokat State Hospital
Other Study IDs: 123456
Record Dates: First submitted 2019-01-26; First posted 2019-01-31 (Actual); Results first posted 2020-04-07 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia Syndrome, Ferritin, Sleep
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fibromyalgia: Non-anemic FMS patients who were diagnosed based on 2011 FMS diagnostic criteria of the American Rheumatology College
- Control: Non-anemic women without a FMS diagnosis

SUMMARY:
The aim of the present study was to evaluate the association between ferritin levels and clinical parameters in patients with fibromyalgia syndrome.

DETAILED DESCRIPTION:
This sectional study included 100 patients with non-anemic FMS diagnosis and 100 patients with non anemic non FMS diagnosis whose ferritin levels were measured within the last four weeks. The participants were evaluated using Fibromyalgia Impact Questionnaire (FIQ), Beck Anxiety Inventory (BAI), Beck Depression Inventory (BDI) and Pittsburg Sleep Quality Index (PSQI) as well as with a questionnaire form about descriptive characteristics. Serum ferritin level of <30 ng/mL was considered iron deficiency.

ELIGIBILITY:
Inclusion Criteria:

* Fibromyalgi syndrome patients
* ferritin levels were measured within the last four weeks

Exclusion Criteria:

* parenteral or enteral iron usage in last four weeks
* hemoglobin level was less than 12 g/dl
* infection
* malignity
* active inflammatory arthritis
* serious skin variations
* serious peripheral vascular disease
* iron storing disorder
* pregnant or lactating patients

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This sectional study included 100 female patients older than 18 years of age who presented to Physical Treatment and Rehabilitation polyclinic in 2016-17 period.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2019-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: sevil okan, Principal Investigator — Doctor

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Fibromiyalgia: 100 Fibromyalgia Patient Group
- Control: 100 Control Group
Period: Overall Study
Arm/Group | Fibromiyalgia | Control
Started | 100 | 100
Completed | 100 | 100
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fibromiyalgia | Control | Total
Number analyzed (Participants) | 100 | 100 | 200
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 100 | 100 | 200
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100 | 100 | 200
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Turkey | 100 | 100 | 200
ferritin level [Median (Inter-Quartile Range); unit: ng/ml] | 20.95 [11.75 to 39.55] | 34.91 [17.87 to 55.12] | 32.92 [14.65 to 47.35]

OUTCOME MEASURES:

1. Primary Outcome: Pitsburgh Sleep Quality Index
Description: Pittsburgh Sleep Quality Index (PSQI) is an 18-item questionnaire measuring sleep quality and disorders in a time period of one month. PSQI measures subjective sleep quality, duration and latency of sleep, sleep disorders, habitual sleep efficiency, daytime dysfunction and use of medication for sleeping. PSQI distinguishes "poor" sleep from "good" sleep.
  minimum score 1 maximum score 9
  ≥5 total points in PSQI mean "poor" sleep. <5 total points in PSQI mean good sleep.
Time Frame: 1 year
Population: 100 This index applied only Firomyalgia syndrome group
Measure: Mean (Standard Deviation); unit: score on a questionnarie
Groups:
- Fibromyalgia: Fibromyalgia syndrome group
Arm/Group | Fibromyalgia
Number analyzed (Participants) | 100
score on a questionnarie | 8.3 (3.77)

2. Primary Outcome: Ferritin Level
Description: Iron deficiency marker
Time Frame: 1 year
Population: 200
Measure: Median (Inter-Quartile Range); unit: ng/ml
Groups:
- Control: Control Group
- Fibromyalgia: Fibromyalgia syndrome
Arm/Group | Control | Fibromyalgia
Number analyzed (Participants) | 100 | 100
ng/ml | 34.91 [17.87 to 55.12] | 20.95 [11.75 to 39.55]

3. Secondary Outcome: Fibromyalgia Impact Questionnarie Scores
Description: Fibromyalgia Impact Questionnaire (FIQ) is a 10-item evaluation tool developed to measure status, prognosis and outcomes of FMS patients. Total points vary from 0 to 100. Higher points show the effect of FMS on functionality.
  mimimum score 0 maximum score 100 higher scores shows poor functionality.
Time Frame: 1 year
Population: 100 This questionnarie applied only Firomyalgia syndrome group
Measure: Mean (Standard Deviation); unit: score on a questionnarie
Groups:
- Fibromiyalgia: 100 Fibromyalgia Patient Group 100 Control Group
Arm/Group | Fibromiyalgia
Number analyzed (Participants) | 100
score on a questionnarie | 61.69 (17.31)

4. Secondary Outcome: Beck Depression Inventory
Description: Beck Depression Inventory (BDI) is a 21-item questionnaire evaluating the presence and severity of depression. Higher points mean heavier depression (0-9 points: minimum depression; 10-18 points: slight depression; 19-29 points: moderate depression; 30-63 points: severe depression).
  minimum 0 maximum 63 points higher scores mean worse outcome.
Time Frame: 1 year
Population: 100 This questionnarie applied only Firomyalgia syndrome group
Measure: Mean (Standard Deviation); unit: score on a questionnarie
Arm/Group | Fibromiyalgia
Number analyzed (Participants) | 100
score on a questionnarie | 15.73 (9.76)

5. Secondary Outcome: Beck Anxiety Inventory
Description: Beck Anxiety Inventory is a short, easily applied and graded, 21-item questionnaire to evaluate the severity of patients' anxiety. Total points vary from 0 to 63 (0-9 points: normal; 10-18 points: slight to moderate anxiety; 19-29 points: moderate to severe anxiety and 30-63 points: very severe anxiety).
  minimum 0 maximum 63 points higher scores mean worse outcome
Time Frame: 1 year
Population: 100 This inventory applied only Firomyalgia syndrome group
Measure: Mean (Standard Deviation); unit: score on a questionnarie
Arm/Group | Fibromiyalgia
Number analyzed (Participants) | 100
score on a questionnarie | 22.58 (11.14)

ADVERSE EVENTS:
Time Frame: no advers event 1 year
Description: no advers event
Arm/Group | Fibromiyalgia | Control
All-Cause Mortality (participants affected / at risk) | 0/100 | 0/100
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/100
Other Adverse Events (participants affected / at risk) | 0/100 | 0/100

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-01): https://cdn.clinicaltrials.gov/large-docs/93/NCT03825393/Prot_SAP_000.pdf